CLINICAL TRIAL: NCT06322550
Title: Influence of Role-expectancy on Patient Reported Outcomes Among Patients With Migraine: a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: beingapatient
Record Dates: First submitted 2024-03-13; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Role-expectancy on Patient Reported Outcomes
Keywords: migraine; role expectation; outcomes; social role; response bias; subjective pain reporting
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Monocenter, randomized, double blind, three-armed clinical trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Migraine Patient (Experimental): 122 migraine patients assigned the role of "patient"
  Interventions: Behavioral: cover story
- Migraine Healthy (Experimental): 122 migraine patients assigned the role of "healthy participant"
  Interventions: Behavioral: cover story
- headache-free controls (No Intervention): 122 headache-free controls with no cover story

INTERVENTIONS:
Behavioral: cover story — After agreeing to participate, migraine patients were randomly given the briefing information and therefore their group allocation. Patients received the cover stories via the allocated flyer with study information and also by the physician from the outpatient clinic. Fifty percent of patients (Migraine as Patients [MP]) received the information that they will take part in a migraine study (compared to healthy controls) and that this study would investigates migraine associated dizziness by watching a visual stimulus (roller coaster video). The protocol for the intervention was standardized and identical for all participants. The other 50% (Migraine as Healthy [MH]) received the information that this study was in cooperation with the University's vertigo Department and that they will take part as controls since they were healthy apart from their migraine.
  Arms: Migraine Healthy; Migraine Patient

SUMMARY:
This study was preregistered 2019 under https://osf.io/nczhj. Since JAMA requires a registration with ClinicalTrials.gov, we post-register the study here with the identical informations from OSF (see there)

Migraine is frequently associated with motion sickness, vestibular symptoms, and abnormal motion and visual processing. Clinical symptoms and underlying brain mechanisms during self-motion visual stimulation were not yet investigated in this population. Therefore the aim is to investigate the behavioral responses from a visually simulated roller coaster ride of patients with migraine and headache-free controls. In order to verify the effect of response bias, part of the patients with migraine will be informed that the study aims to investigate vestibular disorders instead of headache disorders and that they are invited as healthy controls.

DETAILED DESCRIPTION:
We have a three group randomized controlled design. Migraine patients from the headache outpatient clinic will randomly be assigned to get two different cover stories via a flyer with study information and through the physician from the outpatient clinic: 50% of patients will receive the information that they will take part to investigate migraine (by watching the visual stimulus (roller coaster video)). The other 50% will receive the information that they will take part as healthy controls for a headache unrelated study (by watching the visual stimulus (roller coaster video)). Sex and age matched healthy controls will take part in the same experiment and get no additional information but that we investigate the perception of a visual stimulus (roller coaster video). The protocol for the intervention is standardized and identical for all participants.

Migraine patients will be randomly given the priming information and therefore their group allocation. Physicians will allocate by pulling from a randomized equally sized stock of flyers (of which 50% inform for healthy controls and 50% for migraine patients).

Migraine Patients for both migraine groups will be recruited and diagnosed by a neurologist from the UKE headache outpatient clinic. Healthy controls will be recruited via an internet platform for job advertisement. Participants will be paid 10€ for participation. Participants must be at least 18 years old and have signed the informed consent. They are excluded if they have 1. History of any neurological disease, 2. Self-report of diagnosis of vestibular disease, 3. History of trauma or pathology of the cervical spine (e.g., whiplash associated disorder), 4. Pregnancy, 5. Other relevant musculoskeletal, systemic or psychiatric disease.

ELIGIBILITY:
Inclusion Criteria:

* migraine patients following ICHD-3 criteria
* headache free controls

Exclusion Criteria:

* any other headache or pain disorder
* known somatic or psychiatric disorder
* pregnacy or breast feeding
* known vestibular disorder or whiplash injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 366 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
self-reported vestibular symptoms | 1 time point: study day1
  Patients were encouraged to describe their symptoms according to the Barany's Classification of Vestibular Disorders including its form (internal/external vertigo, dizziness or postural symptoms). Outcome was frequency of occurence of vestibular symptoms classified according to the Barany's Classification.

SECONDARY OUTCOMES:
differences in motion sickness susceptibility using a standardized motion sickness questionnaire | 1 time point: study day1
  Motion sickness susceptibility was tested using the MSSQ- short version questionnaire. The outcome is a sum score.
differences in disability level using a standardized motion sickness questionnaire | 1 time point: study day1
  The disability level related to vestibular symptoms was assessed using the Dizziness Handicap Inventory (DHI-G). The outcome is a sum score.
differences in headache days per month | 1 time point: study day1
  The self-report of headache frequency/month was tested.
differences in headache burden and migraine disability questionnaires | 1 time point: study day1
  All participants filled out a questionnaire (migraine disability assessment score - MIDAS) The outcome is a sum-score

CONTACTS AND LOCATIONS:
Overall Officials: Hauke Basedau, MD, Principal Investigator — University Clinic Hamburg
Locations (1):
- UKE, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Researchers meeting the criteria for access to confidential data may access the data upon request, involving the documentation of data access
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: once study is published
Access Criteria: researchers of govermental funded Universities (no commercial companies)

REFERENCES:
- [Derived] May A, Carvalho GF, Schwarz A, Basedau H. Influence of Role Expectancy on Patient-Reported Outcomes Among Patients With Migraine: A Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e243223. doi: 10.1001/jamanetworkopen.2024.3223. PMID 38656579